CLINICAL TRIAL: NCT05559840
Title: S-Condom Uterine Tamponade Using Air Media in Controlling Atraumatic Postpartum Haemorrhage (PPH) - a Randomized Control Trial (RCT)
Brief Title: S-Condom Uterine Tamponade in Controlling Atraumatic Postpartum Haemorrhage (PPH) - RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mamms Institute of Fistula and Womens Health (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Sayeba Akhter, Professor, Mamms Institute of Fistula and Womens Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CMC/PG/2017/39
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Post Partum Hemorrhage
Keywords: Randomised controlled trial, S-condom, postpartum haemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Intervention Model Description: Two treatment strategies will be compared in this pilot study. When PPH will be diagnosed, women will receive standard treatment, 10 units of oxytocin, uterine massage and aortic compression. If bleeding continue, the control group (Group I) will be treated with condom catheter tamponade by inflating the condom with saline according to national protocol. In case of study group (Group II) the condom will be inflated with air.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): The control group (Group I) will be treated with condom catheter tamponade by inflating the condom with saline according to national protocol.
  Interventions: Device: S-Condom Uterine Tamponade
- Group II (Experimental): The study group (Group II) will receive condom catheter that will be inflated with air
  Interventions: Device: Traditional condom catheter

INTERVENTIONS:
Device: S-Condom Uterine Tamponade — The condom catheter will be inflated with air
  Arms: Group I
Device: Traditional condom catheter — The condom catheter will be inflated with saline following national protocol
  Arms: Group II

SUMMARY:
A Randomized Controlled Non inferiority Trial will be conducted to see the feasibility, acceptability and efficacy of S-Condom Uterine Tamponade in women with atraumatic PPH and not responding to first line of treatment.

DETAILED DESCRIPTION:
A Randomized Controlled Non inferiority Trial will be conducted to see the feasibility, acceptability and efficacy of S-Condom Uterine Tamponade in women with atraumatic PPH and not responding to first line of treatment. The women will be divided randomly into two groups, in both groups two condom tied on a catheter will be introduced inside the uterus. In one group (Control group), condom will be inflated with saline and in another group(study group) it will be inflated with air. Time required to stop bleeding will be measured for comparison. Data collected will be analyzed using a quantitative approach and the results will be presented in tables and graphs. If air media proved feasible, acceptable and effective the PPH management will be easier, cost-effective can make a great impact in reaching the target for reduction of maternal mortality in Bangladesh and other resource poor settings.

ELIGIBILITY:
Inclusion Criteria:

* All women who presented with atraumatic postpartum hemorrhage, refractory to first-line treatment (uterine massage and oxytocin) and who will give their consent will be included in the study and will be randomized

Exclusion Criteria:

* Women known to have allergy to latex, or presenting with clinical chorioamnionitis or primary hemorrhage caused by cervical-vaginal lacerations, a uterine rupture, or a placenta accreta will be excluded.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Study participants are all pregnant women with post-partum haemorrhage.
Enrollment: 82 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Time required to stop bleeding | 2 years
  Comparison of the average time to stop bleeding following the intervention and the control

CONTACTS AND LOCATIONS:
Overall Officials: Sayeba Akhter, Dr., Principal Investigator — Mamms Institute of Fistula and Womens Health

IPD SHARING:
Plan to Share IPD: No
We will not share individual participant data with other researchers. We will remove all personal identifier after assigning unique ids to each participant before data entry